CLINICAL TRIAL: NCT03339414
Title: Blood microRNA Depression Change After DHCA
Status: Completed | Type: Observational
Sponsor: China International Neuroscience Institution (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-026283-1
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: collect blood — collect blood at different time point

SUMMARY:
Collect the blood sample per-operation experience deep hypothermia cardiac arrest for aorta artery replacement surgery Collect the blood from the CPB machine and from intravenous injection tube which already set at different time point.

DETAILED DESCRIPTION:
Collect the blood sample per-operation experience deep hypothermia cardiac arrest for aorta artery replacement surgery Collect the blood from the CPB machine and from intravenous injection tube which already set at different time point Test the blood sample of DHCA, analysis the correlation between miR-194 and temperature.

ELIGIBILITY:
Inclusion Criteria:

* aortic dissection patients

Exclusion Criteria:

* other organ disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20-100
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-20 (Actual)

PRIMARY OUTCOMES:
microRNA express change | 1 day
  target microRNA expression change

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohua Wang, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No